CLINICAL TRIAL: NCT00220142
Title: Molecular Markers of Prognosis in Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2348
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To correlate the molecular profile of a series of defined CRCs with prognosis and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* All patients participating in the RMHNHST study of infusional versus bolus 5FU (Saini et al. 2003).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GI unit Royal Marsden Hospital NHS trust (RMHNHST) has co-ordinated and published results from a large multicentre randomised clinical trial of patients with locally advanced CRC (Saini et al. 2003). A total of 716 patients Dukes' B and C CRC operated with curative intent were randomised to receive either bolus or infusional 5FU regimes. Patients treated at the RMHNHST made up the majority of the total sample cohort (n=550). Analysis of results after a median of 19.8 months follow-up showed that infused 5-FU given over 12 weeks resulted in similar survival to bolus 5-FU and FA over a six-month period (log rank p=0.764). There was, however, significantly less toxicity associated with the infusional regime.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2003-11

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom